CLINICAL TRIAL: NCT03037827
Title: Three Different Regimens of Endovenous Laser Ablation With Equal Linear Endovenous Energy Density (The SLEDGE Study): a Prospective, Randomized Multicenter Trial
Brief Title: The Effect of Laser Power and Fiber Traction Speed on the Outcomes of Endovenous Laser Ablation
Acronym: SLEDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinic of Phlebology and Laser Surgery, Chelyabinsk, Russia (Other)
Collaborators: Medalp Private Surgery Clinic (Other); Garantclinic (Other)
Responsible Party: Principal Investigator, Denis Borsuk, Chief surgeon, Clinic of Phlebology and Laser Surgery, Chelyabinsk, Russia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A001
Record Dates: First submitted 2017-01-29; First posted 2017-01-31 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Varicose Veins
Keywords: endovenous laser ablation; radial fiber; linear endovenous energy density; 1470 nm; occlusion rate
MeSH Terms: conditions — Varicose Veins | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endovenous laser ablation (EVLA) 5W (Active Comparator): One of three different regimens of endovenous laser ablation, the fiber pullback speed 0.7 mm/s, laser power 5 W, LEED 71 J/cm
  Interventions: Procedure: Endovenous laser ablation (EVLA); Device: Laser
- Endovenous laser ablation (EVLA) 7W (Active Comparator): One of three different regimens of endovenous laser ablation, the fiber pullback speed 1 mm/s, laser power 7 W, LEED 70 J/cm
  Interventions: Procedure: Endovenous laser ablation (EVLA); Device: Laser
- Endovenous laser ablation (EVLA) 10W (Active Comparator): One of three different regimens of endovenous laser ablation, the fiber pullback speed 1.5 mm/s, laser power 10 W, LEED 67 J/cm
  Interventions: Procedure: Endovenous laser ablation (EVLA); Device: Laser

INTERVENTIONS:
Procedure: Endovenous laser ablation (EVLA) — Endovenous laser ablation with laser wavelength 1470 nm and radial laser fiber
Device: Laser — Device for endovenous laser ablation manufactured by Biolitec AG company (ELVeS system) - diode laser with a wavelength of 1470 nm

SUMMARY:
A multicenter clinical randomized controlled trial, comparing of three different regimens of endovenous laser ablation with equal linear endovenous energy density in patients with insufficiency of the great saphenous vein (GSV). The linear endovenous energy density (LEED) is the main value for standardization EVLA. From many studies, it is known the optimum value of the LEED. However, the same LEED may be obtained by varying the ratio between the laser power and the fiber pullback speed. Power decrease can allow to reduce the incidence of adverse effects of endovenous laser ablation, but keep high efficiency.

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years old Insufficiency of the GSV measured with ultrasound imaging, reflux > 0.5 sec No prior treatment of the insufficient GSV Informed consent

Exclusion Criteria:

Acute deep or superficial vein thrombosis Agenesis of deep vein system Vascular malformation or syndrome Post-thrombotic syndrome, occlusive type Pregnancy Phlebectomy on the thigh Immobility Allergy to lidocaine Arterial insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
The number of participants with a fully obliterated target vein | 3 month
  An ultrasound investigation of the treated vein to find out is the treated vein is fully obliterated or not, and to find out is there any pathological reflux in the vein.

SECONDARY OUTCOMES:
Pain score | day 1
  Pain (numeric rating scale)
Pain score | day 7
  Pain (numeric rating scale)

OTHER OUTCOMES:
Number of patients with adverse events | 3 month
Paresthesia | 3 month
Deep venous thrombosis | day 7
Superficial venous thrombosis | day 7

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Clinic of Phlebology and Laser Surgery, Chelyabinsk
  - GarantClinic, Moscow

IPD SHARING:
Plan to Share IPD: Yes
Data collection will take place at the Russian Registry of Treatment of Chronic Venous Diseases (RRT CVD). Access to the data will be available after completion of the study. To access the data will need to send a request to RRT CVD administrator. Register in Russian. Registry now listed in the database ClinicalTrials.gov, ID NCT03035747 (see references)

REFERENCES:
- [Derived] Borsuk DA, Fokin AA, Lobastov KV, Tauraginskii RA, Zhdanov KO, Zolotov AV, Arkhipov IS, Galchenko MI. A randomized clinical trial to assess the impact of laser power with constant linear endovenous energy density on outcomes of endovenous laser ablation (SLEDGE trial). J Vasc Surg Venous Lymphat Disord. 2023 Sep;11(5):946-953. doi: 10.1016/j.jvsv.2023.03.020. Epub 2023 May 11. PMID 37172934
- See also: the Russian Registry of Treatment of Chronic Venous Diseases (RRT CVD). ClinicalTrials.gov ID: NCT03035747 — http://www.venousregistry.org/